CLINICAL TRIAL: NCT01233596
Title: Monocanalicular Versus Bicanalicular Intubation in the Treatment of Congenital Nasolacrimal Duct Obstruction
Acronym: MCI_vs_BCI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORL-FNO-2010
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Nasolacrimal Duct Obstruction
Keywords: congenital nasolacrimal duct obstruction; monocanalicular intubation; bicanalicular intubation; complications
MeSH Terms: conditions — Lacrimal Duct Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monocanalicular intubation (Active Comparator): Monocanalicular intubations (MCI; n=35 eyes) through the inferior canaliculus intubations performed under general anaeshesia in children between 10 and 36 months of age suffering from congenital nasolacrimal duct obstruction (CNLDO).
  Interventions: Device: Canalicular intubation
- Bicanalicular intubation (Active Comparator): Bicanalicular intubation (BCI; n=35 eyes) performed under general anaeshesia in children between 10 and 36 months of age suffering from congenital nasolacrimal duct obstruction (CNLDO).
  Interventions: Device: Canalicular intubation

INTERVENTIONS:
Device: Canalicular intubation — Intubation through the inferior canaliculus performed under general anaeshesia. The tubes were removed 3-4 months after the tube placement.
  Other Names: silicone tube

SUMMARY:
The aim of the study was to compare the success rate of monocanalicular intubation versus bicanalicular silicone intubation in congenital nasolacrimal duct obstruction in children aged between 10 and 36 months.

DETAILED DESCRIPTION:
In a prospective, nonrandomized comparative study, the monocanalicular intubations (MCI; n=35 eyes) through the inferior canaliculus or bicanalicular intubations (BCI; n=35 eyes) were performed under general anaeshesia in children between 10 and 36 months of age suffering from congenital nasolacrimal duct obstruction (CNLDO). The tubes were removed 3-4 months after the tube placement. Thereafter, the children were followed up for 6 months after the removal of tubes. The therapeutic success was defined as the fluorescein dye disappearance test grade 0-1 corresponding with a complete resolution of previous symptoms. The partial success was defined as improvement with some residual symptoms.

The complete and partial improvement was achieved in 31/35(88.57%) in group I with BCI and in 34/35 (97.14%) in group II with MCI, respectively, and it was not significantly higher (p=0,584).

Complications occurred in both groups. Dislodgement of the tube and premature removal was observed in four cases in group I (BCI), the loss of the tube was observed twice in group II with MCI.. Canalicular slitting was observed in 5 eyes in the group with BCI. Granuloma pyogenicum observed in 2 cases with MCI revealed in a few weeks after the tube removal. Corneal erosion in the inferior medial quadrant was observed in 1 eye with MCI and revealed in a few days after the local treatment without tube removal.

Conclusions: Both MCI and the BCI are effective methods how to treat CNLDO. The advantage of the MCI shows the lower incidence of the canalicular slit and easy placement.

ELIGIBILITY:
Inclusion Criteria:

* congenital nasolacrimal duct obstruction (CNLDO)
* resistance to a conservative therapy and/or probing

Exclusion Criteria:

- children younger than 10 months of age

Ages: 10 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2006-01; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Success rate and complications of monocanalicular and bicanalicular intubation in children | 6 months
  35 consecutive cases of bicanalicular intubations (group I) followed by 35 consecutive cases of monocanalicular intubations (group II). Silicone tubes were removed 3 to 4 months after the surgery. The children were followed up for 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Kominek, MD,PhD,MBA, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czech Republic, Czechia